CLINICAL TRIAL: NCT05569720
Title: First in Human Clinical Trial to Compare Safety and Tolerability Between Intravenous Infusions and Bolus Intravenous Inhection of ApTOLL in Healthy Volunteers
Brief Title: First in Human Study to Compare Safety Between Intravenous Bolus Versus Infusion of ApTOLL
Acronym: APTABOLUS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: aptaTargets S.L. (Industry)
Collaborators: Centro para el Desarrollo Tecnológico Industrial (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APTABOLUS
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — TLR4 antagonist ApTOLL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ApTOLL treatment (Experimental): Volunteers will receive a dose of ApTOLL of 0.1mg/kg administered intravenously as slow infusion one day and as a single bolus intravenous injection the second day. In a third and last admission day, volunteers will receive a dose of ApTOLL of 0.2mg/kg administered as a single bolus intravenous injection.
  Interventions: Drug: ApTOLL

INTERVENTIONS:
Drug: ApTOLL — ApTOLL will be administered as follows:
  * Day 1: a dose of 0.1mg/kg will be administered intravenously as a slow infusion.
  * Day 2: a dose of 0.1mg/kg will be administered intravenously as single bolus injection.
  * Day 3: a dose of 0.2mg/kg will be administered intravenously as single bolus injection.

SUMMARY:
The main objective of the study is to assess the tolerability and safety of ApTOLL administration when comparing intravenous infusion vs. bolus intravenous injection, in healthy volunteers. Pharmacokinetic profile of ApTOLL will be also analysed as secondary objective of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (with no possibility to become pregnant (hysterectomized or menopausal women)) subjects who give their written consent to participate in the study.
* Aged from 18 to 55.
* No clinically significant organic or psychic conditions.
* No clinically significant abnormalities in medical records and physical examination.
* No clinically significant abnormalities in haematology, coagulation, biochemistry, serology and urinalysis .
* No clinically significant abnormalities in vital signs and electrocardiogram.

Exclusion Criteria:

* Subjects affected by an organic or psychic condition.
* Subjects who have received prescribed pharmacological treatment in the last 15 days or any kind of medication in the 48 hours prior to receiving the study medication
* Subjects with body mass index (weight (kg)/height2 (m2)) outside the 18.5-30.0 range.
* History of sensitivity to any drug.
* Positive drug screening (for cannabis, opiates, cocaine and amphetamines).
* Smoker.
* Daily consumers of alcohol and/or acute alcohol poisoning in the last week.
* Having donated blood in the last month before start of the study.
* Participation in another study with administration of investigational drugs in the previous 3 months (if the study was conducted with drug substances marketed in Spain, a period of at least 1 month or 5 half lives, what is longer, will be considered).
* Inability to follow the instructions or collaborate during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Adverse Events | day 1 to day 28
  To evaluate the safety and tolerability between different ways of ApTOLL administration: intravenous infusion versus bolus intravenous injection, and pharmacokinetic characteristics of ApTOLL in healthy volunteers after single dose administration in fasting conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Macarena Hernández, PhD, Study Director — aptaTargets S.L.; Dolores Ochoa, MD, PhD, Principal Investigator — Hospital Universitario La Princesa
Locations (1):
- Clinical Pharmacology Department. Hospital Universitario de La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We have not planned this point yet

REFERENCES:
- [Background] Hernandez-Jimenez M, Martin-Vilchez S, Ochoa D, Mejia-Abril G, Roman M, Camargo-Mamani P, Luquero-Bueno S, Jilma B, Moro MA, Fernandez G, Pineiro D, Ribo M, Gonzalez VM, Lizasoain I, Abad-Santos F. First-in-human phase I clinical trial of a TLR4-binding DNA aptamer, ApTOLL: Safety and pharmacokinetics in healthy volunteers. Mol Ther Nucleic Acids. 2022 Mar 9;28:124-135. doi: 10.1016/j.omtn.2022.03.005. eCollection 2022 Jun 14. PMID 35402075
- [Background] Fernandez G, Moraga A, Cuartero MI, Garcia-Culebras A, Pena-Martinez C, Pradillo JM, Hernandez-Jimenez M, Sacristan S, Ayuso MI, Gonzalo-Gobernado R, Fernandez-Lopez D, Martin ME, Moro MA, Gonzalez VM, Lizasoain I. TLR4-Binding DNA Aptamers Show a Protective Effect against Acute Stroke in Animal Models. Mol Ther. 2018 Aug 1;26(8):2047-2059. doi: 10.1016/j.ymthe.2018.05.019. Epub 2018 Jun 15. PMID 29910175
- [Derived] Hernandez-Jimenez M, Martin-Vilchez S, Mejia-Abril G, Roman M, Luquero-Bueno S, Pineiro D, Ribo M, Abad-Santos F, Ochoa D. Clinical trial to compare safety and tolerability between intravenous infusion and bolus intravenous injection of ApTOLL in healthy volunteers. Mol Ther Nucleic Acids. 2024 Dec 21;36(1):102435. doi: 10.1016/j.omtn.2024.102435. eCollection 2025 Mar 11. PMID 39897575